CLINICAL TRIAL: NCT00934453
Title: A Phase I, Randomized Study to Evaluate the Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) in Healthy Volunteers
Brief Title: Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Global Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 8996
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Healthy adult volunteers; Lactobacillus rhamnosus GG; probiotic; dietary supplement; safety; Safety Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG (Experimental): Lactobacillus rhamnosus GG (LGG) capsules containing 1x10^10 LGG per capsule will be given to volunteers with verbal and written instructions at the baseline visit. Capsules are to be taken orally twice a day dissolved in cow's milk or soy milk on an outpatient basis.
  Interventions: Biological: Lactobacillus rhamnosus GG ATCC 53103
- Placebo (Placebo Comparator): Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day dissolved in cow's milk or soy milk on an outpatient basis.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus rhamnosus GG ATCC 53103 — Study drug capsules (1x10^10 LGG/capsule) are to be taken orally twice a day every day dissolved in cow's milk or soy milk on an outpatient basis for six months.
  Other Names: Culturelle; LGG
  Arms: LGG
Biological: Placebo — Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day dissolved in cow's milk or soy milk on an outpatient basis for six months.
  Arms: Placebo

SUMMARY:
This study is a single site, Phase I, masked, randomized study to evaluate the safety and tolerability of twice daily dosing of LGG (Lactobacillus GG ATCC 53103) in normal healthy adult volunteers. Study drug capsules (1x10^10 LGG/capsule or placebo) will be taken by mouth twice a day with cow's milk or soy milk on an outpatient basis. Volunteers will have study visits at baseline, 1 month, 3 months, 6 months, 7 months, and 12 months where they will be asked about any medical problems that have come up since the last study visit, have vital signs taken, review current medication use, and review any signs of potential adverse events. Blood and urine samples will also be collected at these visits, as well as throat and stool samples.

Our goal is to assess the safety and tolerability of LGG when administered to healthy adult volunteers twice a day. Assessment of safety will be determined by vital sign measurements, physical examinations, clinical laboratory tests, and from the incidence and severity of adverse events that occur during study participation. Additionally, we will assess whether LGG colonizes the throat and/or gastrointestinal tract of healthy adult volunteers and assess the effect of LGG on the bacteria that normally live in the throat and GI tract by using culture-independent techniques. Volunteers enrolled in this study will also be invited to participate in a companion genetic study that will investigate the host immune response to the bacteria in LGG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years, inclusive.
* Expressed interest and ability to fulfill the study requirements.
* Be in general good health as determined by a screening evaluation within 30 days of the first dose of LGG or placebo.
* Able to ingest the study drug (LGG or placebo) dissolved in a small amount of cow's milk or soy milk orally (no feeding tube).
* Willing to prevent pregnancy - Women must agree not to become pregnant or breastfeed from the time of study enrollment until at least 3 months after the last dose of study drug. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to practice an acceptable method of birth control, such as hormonal or barrier birth control. A woman is eligible if she is monogamous with a vasectomized male. Sexually active male volunteers without vasectomy must agree to use a barrier method of contraception for 3 months after the last dose of study drug.
* Willing to comply with protocol and report on compliance and side effects during study period.
* Informed consent obtained and signed prior to screening.

Exclusion Criteria:

* Consumption of supplements or food products containing LGG or probiotics 30 days prior to the start of the study or consumption of yogurt that has "live and active cultures" seal.
* Known or suspected allergies to probiotics, Lactobacillus, microcrystalline cellulose, gelatin, or any antibiotic that may be used to treat LGG bacteremia or infection (Ampicillin, Clindamycin, Moxifloxacin).
* Received oral or parenteral antibiotics within 4 weeks of enrollment or prescribed antibiotics on day of enrollment.
* Drug or alcohol abuse within previous 12 months.
* Major surgery or endoscopy within last 3 months.
* Daily prescription or over-the-counter medicines except for vitamins, birth control products, and hormone replacement therapy.
* Presence of any of the following:

  * Abnormal vital signs or clinically significant physical findings such as murmur (other than functional), hepatosplenomegaly, jaundice, lymphadenopathy, or focal neurological deficit
  * Indwelling catheter or implanted hardware/prosthetic device or feeding tube
  * Febrile illness (oral temperature >37 degrees Celsius) or one or more episodes of diarrhea within 72 hours of baseline visit (first dose of study drug)
  * Active bowel leak, acute abdomen, colitis, or active GI disease or history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, or inflammatory bowel disease
  * History of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease
  * Underlying structural heart disease or previous history of endocarditis or valve replacement
  * Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy, neutrophil count <500/mm^3, or an anticipated drop in the neutrophil count to <500/mm3
  * History of cancer
  * History of collagen vascular disease
  * Active TB
* Women only - pregnant, planning on becoming pregnant within the next 9 months, breastfeeding, positive urine pregnancy test during screening or within 24 hours of first dose of study drug, or unwilling to undergo pregnancy testing.
* Positive drug or alcohol testing at screening or within 24 hours of first dose of study drug, or unwilling to undergo drug and alcohol testing.
* Screening laboratory tests greater than upper normal limit (ULN) or less than lower normal limit (LLN):

  * White blood cell <LLN or >ULN
  * Platelets <LLN
  * Hemoglobin <LLN
  * Creatinine >ULN
  * Blood urea nitrogen >ULN
  * Aspartate aminotransferase >ULN
  * Alanine aminotransferase >ULN
  * Alkaline phosphatase >ULN
  * Bilirubin >ULN
  * Glucose (nonfasting ) >109 mg/dL
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer participating in the study or would make it unlikely the volunteer could complete the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Vital signs, including weight, temperature, resting blood pressure, heart rate, and respiratory rate, will be taken. The rate of notable vital sign abnormalities and changes from baseline to each post-baseline visit will be summarized by group. | Baseline, 1 month, 3 months, 6 months, 7 months, 12 months
Physical examination will be performed. The abnormal findings in physical examination will be summarized by treatment group using descriptive statistics. | Baseline, 1 month, 3 months, 6 months, 7 months, 12 months
Clinical laboratory tests - abnormal values, clinically significant abnormal range, overall lab data, and changes from baseline will be summarized by cohort. | Baseline, 1 month, 3 months, 6 months, 7 months, 12 months
Adverse event assessment | Baseline, day 3, day 7, day 14, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 12 months

SECONDARY OUTCOMES:
Throat samples will be obtained for routine culture including quantitative analyses of LGG and also for extraction of bacterial DNA to describe the microbiota (bacteria normally present) of the oropharynx. | Baseline, month 1, month 3, month 6, month 7, month 12
Stool samples will be obtained for routine culture including quantitative analyses of LGG and also for extraction of bacterial DNA to describe the microbiota (bacteria normally present) of the GI tract. | Baseline, month 1, month 3, month 6, month 7, month 12
Additional blood samples (approximately 1/2 teaspoon per study visit) will be collected to determine the expression of immune associated markers in the blood if volunteers participate in the companion genetic study. | Baseline, month 1, month 3, month 6, month 7 and month 12
Stool samples (already collected - see above) will also be evaluated for changes in intestinal microflora if volunteers participate in the companion genetic study. | Baseline, 1 month, 3 months, 6 months, 7 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts